CLINICAL TRIAL: NCT03026426
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of a Mobile Technology Intervention in the Treatment of Depressive Symptoms in People With Diabetes or Hypertension in Peru
Brief Title: Effectiveness of a mHealth Intervention for the Treatment of Depression in People With Diabetes or Hypertension in Peru
Acronym: LATIN-MHPeru
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: University of Sao Paulo General Hospital (Other); National Institute of Mental Health (NIMH) (NIH); Northwestern University (Other)
Responsible Party: Principal Investigator, Jaime Miranda, Dr., Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U19MH098780-02 Peru; 1U19MH098780 (NIH)
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Depression; Diabetes; Hypertension
Keywords: Depression; Chronic diseases; Mobile technology; Clinical trial
MeSH Terms: conditions — Depression; Diabetes Mellitus; Hypertension; Chronic Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONEMO (Experimental): Participants in the intervention arm will receive a smartphone with CONEMO, an application with 18 sessions that are delivered 3 times a week for 6 weeks.
  Additionally, all study participants, including those in the intervention arm, who present a high risk of suicide and/or have a PHQ-9 score ≥20 are referred to the system for follow up. Participants with lower levels of depressive symptoms receive the recommendation of going to a mental health professional.
  Interventions: Behavioral: CONEMO
- Control Group (No Intervention): Participants in the control group will receive enhanced usual care. Participants who present a high risk of suicide and/or have a PHQ-9 score ≥20 are referred to the system for follow up. Participants with lower levels of depressive symptoms receive the recommendation of going to a mental health professional.

INTERVENTIONS:
Behavioral: CONEMO — Participants will be offered a behavioral activation-based intervention delivered by an application for smartphones (CONEMO) oriented to encourage them to be more active and to incorporate more activities in participants' everyday life.
  Nurses will train participants to use CONEMO, make phone calls when participants are non-adherent, and provide technical support when necessary. Nurses will be supervised by clinical psychologists.
  Arms: CONEMO

SUMMARY:
Background: Depression is a common comorbidity of physical chronic diseases such as diabetes and/or hypertension and constitutes an important public health problem. It correlates negatively with the patients' quality of life and self-care, as well as compliance with medical treatment. In low- and middle-income countries depression often goes unrecognized and untreated, and there are limited human resources to treat depression and other mental problems.

Aim: The present study aims to test a 6-week low-intensity psychological intervention (CONEMO - CONtrol EMOcional) delivered by a smartphone application to people with depressive symptoms and co-morbid diabetes and/or hypertension recruited in primary health care centers and public hospitals in Lima, Peru.

DETAILED DESCRIPTION:
Epidemiologic research has clearly established the significant public health importance of mental disorders in low- and middle-income countries (LMIC). Among mental disorders, depression has become a major problem as a single condition and, more often, as part of complex clinical settings in which multiple conditions and risk factors are combined.

There is substantial co-morbidity between depression and chronic physical conditions, and the outcome of both conditions is impaired when there is this co-morbidity. Most of the disease burden in Latin America is attributable to chronic diseases such as cardio-vascular diseases as hypertension and diabetes, as well as to mental disorders such as depression. Despite the public health impact of depression, it often goes unrecognized and untreated. One important factor for this treatment gap are the limited financial and human resources. The mental health resources available in LMIC are often not optimally distributed either. Funds and trained personnel are typically allocated to tertiary health care services, such as psychiatric hospitals.

Therefore, any short- and medium-term efforts to develop, evaluate, and disseminate effective mental health interventions in LMIC must adapt to these severe workforce shortages, resource limitations, and budgetary inequities. The mental health field needs to consider developing self-help automated interventions that can reach people where there is insufficient access to specialized health care providers. This can be partially addressed applying two strategies: 1) increasing effective self-management; and 2) task-shifting roles to less specialized but appropriately trained health workers.

The investigators are conducting a randomized controlled trial with individuals with chronic diseases, i.e. hypertension and/or diabetes, and symptoms of depression in primary health centers and hospitals in Lima, Peru. Participants will be randomly assigned to the control arm or the intervention arm. The later will receive the CONEMO intervention, monitored by nurses.

The focus of this project is on using a self-help intervention that provides advice, support, and motivation. However, studies suggest that depressed patients left alone with the devices fail to make good use of self-help interventions. Therefore, nurses will monitor participants by a web-based dashboard connected to the smartphone application (CONEMO), motivate to continue using CONEMO if participants are non-adherent and give technical support. Nurses will take part in supervision meetings at least once a week.

Method:

CONEMO is a randomized controlled trial conducted with 432 chronic patients who present diabetes and/or hypertension and depressive symptoms recruited in primary health care centers and public hospitals in Lima, Peru. Half of these participants will be randomized to receive the CONEMO intervention and the other half will receive enhanced usual care. The randomization will be made based on 2 strata: the health center/hospital the participant comes from and his/her PHQ9 score at screening (≤14; ≥15).

The intervention, based on behavior activation, is delivered by a smartphone and monitored by nurses who mediate this intervention, motivating and supporting the participant and monitoring his/her performance. The CONEMO intervention is delivered 3 times a week for a period of 6 weeks, summing up to a total of 18 sessions. Intensity of depressive symptoms is assessed by research assistants using the PHQ-9 at baseline, 3- and 6-month follow-up assessments.

Outcomes:

The primary outcome in this study is the proportion of participants with a reduction of 50% or more in the PHQ-9 score at the 3-month assessment. The secondary outcomes are the proportion of participants with a reduction of 50% or more in the PHQ-9 score at the 6-month assessment, and the improvement in quality of life, adherence to diabetes, level of activity and hypertension medication and social functioning. There will also be a cost-effectiveness evaluation using a intention to treat analysis, and a process evaluation. For the process evaluation, data will be collected from questionnaires about the CONEMO system, filled out by with participants at 3 months after inclusion, and interviews with the nurses at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Presenting depressive symptoms (PHQ9≥10)
* Clinical diagnosis of diabetes and/or hypertension
* Able to read

Exclusion Criteria:

* If pregnant, the diagnosis of hypertension or diabetes is not related to the current pregnancy
* Moderate or severe suicide risk (Level B2 or C measured by S-RAP)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a reduction of 50% or more in the Patient Health Questionnaire (PHQ-9) score at the 3-month assessment | 3 months after inclusion
  Presence and severity of depressive symptoms is measured with the PHQ-9. A reduction of 50% or more in the PHQ-9 score at the 3-month assessment as compared to the PHQ-9 score at baseline will be considered as treatment success.

SECONDARY OUTCOMES:
Proportion of participants with a reduction of 50% or more in the PHQ-9 score at the 6-month assessment | 6 months after inclusion
  Presence and severity of depressive symptoms is measured with the PHQ-9. A reduction of 50% or more in the PHQ-9 score at the 6-month assessment as compared to the PHQ-9 score at baseline will be considered as treatment success.
Improvement in scores for Quality of Life measured by the EQD5 at the 3- and 6-month assessment | 3 and 6 months after inclusion
  Quality of life will be measured at the 3- and 6-month assessments and compared to baseline using the EQ-5D, a standardized instrument that investigates 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Proportion of participants who improve adherence to diabetes or hypertension medications, evaluated by the Morisky questionnaire at the 3- and 6-month assessments | 3 and 6 months after inclusion
  Medication adherence to diabetes or hypertension will be measured using the Morisky Medication Adherence Scale (MMAS-4) at the 3- and 6-month assessments after inclusion and compared to baseline.
Proportion of participants who improve on social functioning at the 3- and 6-month assessments compared to the baseline. | 3 and 6 months after inclusion
  Social functioning will be assessed with the WHO-DAS 2.0 12-item Interviewer-administered version in Spanish at the 3- and 6-month assessments after inclusion and compared to baseline. Its structure is unidimensional and has high internal consistency.
Cost-effectiveness: Number of medical consultations, hospitalizations, and visits to the health care team | 3 and 6 months after inclusion
  Data on the use of health services will be collected at baseline, 3-month and 6-month assessments. Information about medical consultations, hospitalizations, and visits to the health care team will be obtained with a standardized questionnaire and cost-effectiveness analysis will be conducted.
Proportion of participants who improve level of activity at the 3- and 6-month assessments | 3 and 6 months after inclusion
  Level of activity will be evaluated by the short form of the Behavioral Activation for Depression Scale (BADS) and assessed at baseline, 3-month, and 6-month follow-ups. It is a 9-item scale used to measure the frequency of activation and avoidance behaviors hypothetically underlying depression mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Menezes, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital; Ricardo B Araya, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Jaime Miranda, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Lisa Colpe, PhD, Principal Investigator — National Institute of Mental Health (NIMH); Francisco Diez-Canseco, MSc, MPH, Study Chair — Universidad Peruana Cayetano Heredia; Lena R Brandt, MSc, Study Chair — Universidad Peruana Cayetano Heredia
Locations (8):
- Peru (8):
  - Policlínico Bellavista, Callao
  - Policlínico Hermana María Donrose Sutmöller, Callao
  - Hospital Nacional Dos de Mayo, Lima
  - Policlínico Juan José Rodríguez Lazo, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - CAP III Carabayllo, Lima
  - Universidad Peruana Cayetano Heredia, Lima

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Menezess PR, Araya R, Miranda J, Mohr DC, Price le SN. The Latin American treatment and innovation network in mental health h (LATINMH): rationale and scope. Rev Fac Cien Med Univ Nac Cordoba. 2015;72(4):321-30. PMID 27107284
- [Derived] Claro HG, Menezes PR, Fernandes IF, Seward N, Miranda JJ, Saidel MGB, Baquete AGL, Daley KL, Aschar S, Cruz DV, Castro HCM, Rocha T, Quayle J, Peters TJ, Araya R. Do baseline participant characteristics impact the effectiveness of a mobile health intervention for depressive symptoms? A post-hoc subgroup analysis of the CONEMO trials. Braz J Psychiatry. 2024;46:e20233172. doi: 10.47626/1516-4446-2023-3172. Epub 2024 Jan 30. PMID 38345934
- [Derived] Toyama M, Cavero V, Araya R, Menezes PR, Mohr DC, Miranda JJ, Diez-Canseco F. Participants' and Nurses' Experiences With a Digital Intervention for Patients With Depressive Symptoms and Comorbid Hypertension or Diabetes in Peru: Qualitative Post-Randomized Controlled Trial Study. JMIR Hum Factors. 2022 Sep 15;9(3):e35486. doi: 10.2196/35486. PMID 36107482
- [Derived] Vera Cruz Dos Santos D, Coelho de Soarez P, Cavero V, U Rocha TI, Aschar S, Daley KL, Garcia Claro H, Abud Scotton G, Fernandes I, Diez-Canseco F, Brandt LR, Toyama M, Martins Castro HC, Miranda JJ, Araya R, Quayle J, Rossi Menezes P. A Mobile Health Intervention for Patients With Depressive Symptoms: Protocol for an Economic Evaluation Alongside Two Randomized Trials in Brazil and Peru. JMIR Res Protoc. 2021 Oct 13;10(10):e26164. doi: 10.2196/26164. PMID 34643538
- [Derived] Araya R, Menezes PR, Claro HG, Brandt LR, Daley KL, Quayle J, Diez-Canseco F, Peters TJ, Vera Cruz D, Toyama M, Aschar S, Hidalgo-Padilla L, Martins H, Cavero V, Rocha T, Scotton G, de Almeida Lopes IF, Begale M, Mohr DC, Miranda JJ. Effect of a Digital Intervention on Depressive Symptoms in Patients With Comorbid Hypertension or Diabetes in Brazil and Peru: Two Randomized Clinical Trials. JAMA. 2021 May 11;325(18):1852-1862. doi: 10.1001/jama.2021.4348. PMID 33974019
- [Derived] Rocha TIU, Aschar SCAL, Hidalgo-Padilla L, Daley K, Claro HG, Martins Castro HC, Dos Santos DVC, Miranda JJ, Araya R, Menezes PR. Recruitment, training and supervision of nurses and nurse assistants for a task-shifting depression intervention in two RCTs in Brazil and Peru. Hum Resour Health. 2021 Feb 5;19(1):16. doi: 10.1186/s12960-021-00556-5. PMID 33546709